CLINICAL TRIAL: NCT03212950
Title: Day and Night Closed-Loop Glycemic Control With Faster-Acting Insulin Aspart in Young Adults With Type 1 Diabetes Using DreaMed Glucositter - The Fast PHYSI-DREAM Study
Brief Title: Closed-Loop With Faster Aspart in Young Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD-FAST-01
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast-CL (Experimental): Glucose control using DreaMed Glucositter and Fiasp® (Fast-CL)
  Interventions: Drug: Fast-CL
- Regular-CL (Active Comparator): Glucose control using DreaMed Glucositter and regular insulin Aspart
  Interventions: Drug: Regular-CL

INTERVENTIONS:
Drug: Fast-CL — After the admission we will insert new insulin (blinded) into the insulin pump. At 13:00 they will have lunch (with manual bolus). At 15:00 we will start CL control, participants/investigators will not be allowed to deliver manual bolus till the end of the study period. All meals and afternoon exercise (in the time between 16:30 and 19:30) will be unannounced and managed with CL.
  Other Names: Faster Acting Insulin Aspart and DreaMed Glucositter
  Arms: Fast-CL
Drug: Regular-CL — After the admission we will insert new insulin (blinded) into the insulin pump. At 13:00 they will have lunch (with manual bolus). At 15:00 we will start CL control, participants/investigators will not be allowed to deliver manual bolus till the end of the study period. All meals and afternoon exercise (in the time between 16:30 and 19:30) will be unannounced and managed with CL.
  Other Names: Insulin Aspart and DreaMed Glucositer
  Arms: Regular-CL

SUMMARY:
A randomized, double-blinded (for insulin type), single centre, crossover design young adult study, on 20 subjects with type 1 diabetes (T1D), aged 18 to 25 (inclusive) years, measuring time in glucose values within 3.9 - 10 mmol/l (70-180 mg/dl) under supervision of DreaMed Glucositter using either faster-acting insulin Aspart (Fiasp®, European Medicines Agency number EMEA/H/C/004046) or normal acting insulin Aspart.

Study duration will be about 3 weeks per subject, 5 month overall.

The objectives of this clinical investigation is:

1. to evaluate the safety and efficacy of blood glucose control using the DreaMed Glucositter with Fiasp® in young adults with T1D during and after unannounced afternoon physical activity and unannounced meals, in a controlled in-hospital environment.

Primary endpoint is significant between-group difference (intervention Fast-CL versus control Regular-CL) in time within range of glucose values within 3.9 - 10 mmol/l (70-180 mg/dl) during the unannounced afternoon exercise and unannounced standardized meals from 15:00 till 18:00 next day based on sensor glucose readings.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has documented T1D, as defined by the American Diabetes Association and World Health Organization (ADA/WHO) for at least 1 year prior to study enrolment
2. Documented evidence should exist within the patient history of T1D
3. The subject is between 18 and 25 years of age (inclusive) at the time of enrolment
4. The subject has been treated with an insulin pump for at least 3 months
5. The subject has an A1C value ≤ 9% based on analysis from the local laboratory at the time of enrolment

   ● A1C testing must follow National Glycohemoglobin Standardization Program (NGSP) standards.
6. The subject is willing to follow all study instructions
7. Subject is available for the entire study duration and follow-up visits
8. Subject is willing to perform daily self-monitoring of blood glucose (SMBG) and required sensor calibrations
9. If subject has celiac/Hashimoto disease, the disease has to be adequately treated as determined by the investigator
10. Subject has a BMI above 5th centile and below 95th centile for age, respectively.

Exclusion Criteria:

1. Concomitant diseases that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, history of adrenal insufficiency) or other medical conditions, which in the investigator's opinion, may compromise patient safety; Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.
2. Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study (e.g. current treatment for cancer, mental disorder)
3. Subject is taking or has taken oral or parenteral glucocorticoids within 1 month prior to screening, or plans to take oral or parenteral glucocorticoids during the study. Exceptions: Short term oral glucocorticoids up to 7 days, inhaled steroids.
4. Subject is taking antidiabetic agents or other medications, which could be a contraindication to participation in the study by the judgment of the investigator.
5. Subject is participating in another study of a medical device or drug that could affect glucose measurements or glucose management or Receipt of any investigational medical product within 1 month prior to screening (Visit 1).
6. Female subject of child-bearing potential who is pregnant, breast-feeding, or planning to become pregnant during the study.
7. Subject has a history of one or more episodes of Diabetic Ketoacidosis (DKA) requiring hospitalization within a month prior to the screening.
8. Subject has current or recent history of alcohol or drug abuse.
9. Subject has visual impairment or hearing loss, which in the investigator's opinion, may compromise patient ability to perform study procedures safely (child and parent should be evaluated as a unit).

   -

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Time within range 3.9 - 10 mmol/l (70 - 180 mg/dl) | 28 hours
  Primary endpoint is significant between-group difference (intervention Fast-CL versus control Regular-CL) in time within range 3.9 - 10 mmol/l (70 - 180 mg/dl) during the unannounced afternoon exercise and the afternoon/night after (till 18:00 next day) based on sensor glucose readings.

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Prof, MD, Principal Investigator — University of Ljubljana, Faculty of Medicine
Locations (1):
- UMC-University Children's Hospital, Ljubljana, Slovenia

REFERENCES:
- [Background] Quirk H, Blake H, Tennyson R, Randell TL, Glazebrook C. Physical activity interventions in children and young people with Type 1 diabetes mellitus: a systematic review with meta-analysis. Diabet Med. 2014 Oct;31(10):1163-73. doi: 10.1111/dme.12531. PMID 24965376
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Chimen M, Kennedy A, Nirantharakumar K, Pang TT, Andrews R, Narendran P. What are the health benefits of physical activity in type 1 diabetes mellitus? A literature review. Diabetologia. 2012 Mar;55(3):542-51. doi: 10.1007/s00125-011-2403-2. Epub 2011 Dec 22. PMID 22189486
- [Background] Kriska AM, LaPorte RE, Patrick SL, Kuller LH, Orchard TJ. The association of physical activity and diabetic complications in individuals with insulin-dependent diabetes mellitus: the Epidemiology of Diabetes Complications Study--VII. J Clin Epidemiol. 1991;44(11):1207-14. doi: 10.1016/0895-4356(91)90153-z. PMID 1941015
- [Background] Miller RG, Mahajan HD, Costacou T, Sekikawa A, Anderson SJ, Orchard TJ. A Contemporary Estimate of Total Mortality and Cardiovascular Disease Risk in Young Adults With Type 1 Diabetes: The Pittsburgh Epidemiology of Diabetes Complications Study. Diabetes Care. 2016 Dec;39(12):2296-2303. doi: 10.2337/dc16-1162. Epub 2016 Sep 21. PMID 27654986
- [Background] Tsalikian E, Mauras N, Beck RW, Tamborlane WV, Janz KF, Chase HP, Wysocki T, Weinzimer SA, Buckingham BA, Kollman C, Xing D, Ruedy KJ; Diabetes Research In Children Network Direcnet Study Group. Impact of exercise on overnight glycemic control in children with type 1 diabetes mellitus. J Pediatr. 2005 Oct;147(4):528-34. doi: 10.1016/j.jpeds.2005.04.065. PMID 16227041
- [Background] Guelfi KJ, Jones TW, Fournier PA. The decline in blood glucose levels is less with intermittent high-intensity compared with moderate exercise in individuals with type 1 diabetes. Diabetes Care. 2005 Jun;28(6):1289-94. doi: 10.2337/diacare.28.6.1289. PMID 15920041
- [Background] Bussau VA, Ferreira LD, Jones TW, Fournier PA. A 10-s sprint performed prior to moderate-intensity exercise prevents early post-exercise fall in glycaemia in individuals with type 1 diabetes. Diabetologia. 2007 Sep;50(9):1815-1818. doi: 10.1007/s00125-007-0727-8. Epub 2007 Jun 22. PMID 17583795
- [Background] Bussau VA, Ferreira LD, Jones TW, Fournier PA. The 10-s maximal sprint: a novel approach to counter an exercise-mediated fall in glycemia in individuals with type 1 diabetes. Diabetes Care. 2006 Mar;29(3):601-6. doi: 10.2337/diacare.29.03.06.dc05-1764. PMID 16505513
- [Background] Tonoli C, Heyman E, Roelands B, Buyse L, Cheung SS, Berthoin S, Meeusen R. Effects of different types of acute and chronic (training) exercise on glycaemic control in type 1 diabetes mellitus: a meta-analysis. Sports Med. 2012 Dec 1;42(12):1059-80. doi: 10.1007/BF03262312. PMID 23134339
- [Background] Adolfsson P, Nilsson S, Albertsson-Wikland K, Lindblad B. Hormonal response during physical exercise of different intensities in adolescents with type 1 diabetes and healthy controls. Pediatr Diabetes. 2012 Dec;13(8):587-96. doi: 10.1111/j.1399-5448.2012.00889.x. PMID 23173876
- [Background] Robertson K, Riddell MC, Guinhouya BC, Adolfsson P, Hanas R; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Exercise in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:203-23. doi: 10.1111/pedi.12176. No abstract available. PMID 25182315
- [Background] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459
- [Background] Phillip M, Battelino T, Atlas E, Kordonouri O, Bratina N, Miller S, Biester T, Stefanija MA, Muller I, Nimri R, Danne T. Nocturnal glucose control with an artificial pancreas at a diabetes camp. N Engl J Med. 2013 Feb 28;368(9):824-33. doi: 10.1056/NEJMoa1206881. PMID 23445093
- [Background] Anderson SM, Raghinaru D, Pinsker JE, Boscari F, Renard E, Buckingham BA, Nimri R, Doyle FJ 3rd, Brown SA, Keith-Hynes P, Breton MD, Chernavvsky D, Bevier WC, Bradley PK, Bruttomesso D, Del Favero S, Calore R, Cobelli C, Avogaro A, Farret A, Place J, Ly TT, Shanmugham S, Phillip M, Dassau E, Dasanayake IS, Kollman C, Lum JW, Beck RW, Kovatchev B; Control to Range Study Group. Multinational Home Use of Closed-Loop Control Is Safe and Effective. Diabetes Care. 2016 Jul;39(7):1143-50. doi: 10.2337/dc15-2468. Epub 2016 Apr 13. PMID 27208316
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Stewart Z, Cheng P, Kollman C, Acerini CL, Dunger DB, Hovorka R. Day-and-Night Hybrid Closed-Loop Insulin Delivery in Adolescents With Type 1 Diabetes: A Free-Living, Randomized Clinical Trial. Diabetes Care. 2016 Jul;39(7):1168-74. doi: 10.2337/dc15-2078. Epub 2016 Jan 6. PMID 26740634
- [Background] Kovatchev B, Tamborlane WV, Cefalu WT, Cobelli C. The Artificial Pancreas in 2016: A Digital Treatment Ecosystem for Diabetes. Diabetes Care. 2016 Jul;39(7):1123-6. doi: 10.2337/dc16-0824. No abstract available. PMID 27330124
- [Background] Turksoy K, Paulino TM, Zaharieva DP, Yavelberg L, Jamnik V, Riddell MC, Cinar A. Classification of Physical Activity: Information to Artificial Pancreas Control Systems in Real Time. J Diabetes Sci Technol. 2015 Oct 6;9(6):1200-7. doi: 10.1177/1932296815609369. PMID 26443291
- [Background] Taleb N, Emami A, Suppere C, Messier V, Legault L, Ladouceur M, Chiasson JL, Haidar A, Rabasa-Lhoret R. Efficacy of single-hormone and dual-hormone artificial pancreas during continuous and interval exercise in adult patients with type 1 diabetes: randomised controlled crossover trial. Diabetologia. 2016 Dec;59(12):2561-2571. doi: 10.1007/s00125-016-4107-0. Epub 2016 Oct 4. PMID 27704167
- [Background] DeBoer MD, Chernavvsky DR, Topchyan K, Kovatchev BP, Francis GL, Breton MD. Heart rate informed artificial pancreas system enhances glycemic control during exercise in adolescents with T1D. Pediatr Diabetes. 2017 Nov;18(7):540-546. doi: 10.1111/pedi.12454. Epub 2016 Oct 13. PMID 27734563
- [Background] Riddell MC, Zaharieva DP, Yavelberg L, Cinar A, Jamnik VK. Exercise and the Development of the Artificial Pancreas: One of the More Difficult Series of Hurdles. J Diabetes Sci Technol. 2015 Oct 1;9(6):1217-26. doi: 10.1177/1932296815609370. PMID 26428933
- [Background] Heinemann L, Muchmore DB. Ultrafast-acting insulins: state of the art. J Diabetes Sci Technol. 2012 Jul 1;6(4):728-42. doi: 10.1177/193229681200600402. PMID 22920797
- [Background] Heise T, Hovelmann U, Brondsted L, Adrian CL, Nosek L, Haahr H. Faster-acting insulin aspart: earlier onset of appearance and greater early pharmacokinetic and pharmacodynamic effects than insulin aspart. Diabetes Obes Metab. 2015 Jul;17(7):682-8. doi: 10.1111/dom.12468. Epub 2015 May 8. PMID 25846340
- [Background] Bode BW, Johnson JA, Hyveled L, Tamer SC, Demissie M. Improved Postprandial Glycemic Control with Faster-Acting Insulin Aspart in Patients with Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion. Diabetes Technol Ther. 2017 Jan;19(1):25-33. doi: 10.1089/dia.2016.0350. Epub 2017 Jan 5. PMID 28055230
- [Background] Heise T, Zijlstra E, Nosek L, Rikte T, Haahr H. Pharmacological properties of faster-acting insulin aspart vs insulin aspart in patients with type 1 diabetes receiving continuous subcutaneous insulin infusion: A randomized, double-blind, crossover trial. Diabetes Obes Metab. 2017 Feb;19(2):208-215. doi: 10.1111/dom.12803. Epub 2016 Nov 14. PMID 27709762
- [Background] American Diabetes Association. Executive summary: Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S5-13. doi: 10.2337/dc14-S005. No abstract available. PMID 24357214
- [Background] Ly TT, Maahs DM, Rewers A, Dunger D, Oduwole A, Jones TW; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Assessment and management of hypoglycemia in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:180-92. doi: 10.1111/pedi.12174. Epub 2014 Jul 12. No abstract available. PMID 25040141
- [Derived] Dovc K, Piona C, Yesiltepe Mutlu G, Bratina N, Jenko Bizjan B, Lepej D, Nimri R, Atlas E, Muller I, Kordonouri O, Biester T, Danne T, Phillip M, Battelino T. Faster Compared With Standard Insulin Aspart During Day-and-Night Fully Closed-Loop Insulin Therapy in Type 1 Diabetes: A Double-Blind Randomized Crossover Trial. Diabetes Care. 2020 Jan;43(1):29-36. doi: 10.2337/dc19-0895. Epub 2019 Oct 1. PMID 31575640